CLINICAL TRIAL: NCT00167037
Title: Fast Stepping in Stroke Patients for Fall Prediction and Prevention:Control Mechanisms and Clinical Implications
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 56m3
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-09

CONDITIONS: Stroke
Keywords: Hemiplegia; Waist pulling perturbation; Reactive balance strategy; Trajectory of center of pressure; Parameters of center of pressure
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
The purpose of this study was to compare the balance strategy, as well as center of pressure (COP) trajectory and parameters between healthy adults and patients with hemiplegia in response to slow- and fast-speed waist- pulling perturbations in forward, left, right, and backward directions.

DETAILED DESCRIPTION:
The ability to quickly respond to external perturbations is an important capacity of stroke patients to maintain dynamic balance in activities of daily living. The purpose of this study was to compare the balance strategy, as well as center of pressure (COP) trajectory and parameters between healthy adults and patients with hemiplegia in response to slow- and fast-speed waist- pulling perturbations in forward, left, right, and backward directions.

ELIGIBILITY:
Inclusion Criteria:

Healthy adults

* Age ang Sex are correspond with the stroke subjects(between 40 and 75 years old)
* being willing to accept one-year follow-up examination
* being willing to sign an informed consent approved by the Human Subjects Committee of the National Taiwan University Hospital Stroke patients
* between 40 and 75 years old
* stroke confirmed by ICD-10-CM (including I60, I61, I62, I63, I67, and I69)
* first stroke with single side hemiplegia and received acute treatment at NTUH
* being willing to sign an informed consent approved by the Human Subjects Committee of the National Taiwan University Hospital
* able to step forward, laterally and backward independently without assistive device

Excursion criteria:

Healthy adults

* - having other neurological diseases, or moderate to severe neuromuscular or musculoskeletal disorders, or disorders from systematic diseases those would influence the belance or motor ability Stroke patients
* having unstable vital sign, unconsciousness, or obvious cognitive, perception, and language impairment, and couldn't communicate with the experimenters
* having other neurological diseases, or moderate to severe neuromuscular or musculoskeletal or cardiovascular disorders, or disorders from systematic diseases other than stroke

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 1999-08; Study Completion 2002-07

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Fang Tang, PhD, Principal Investigator — National Taiwan University Hospital